CLINICAL TRIAL: NCT03469479
Title: The Efficacy and Safety of Resection Plus Neoadjuvant Hepatic Arterial Infusion Chemotherapy Compared With Resection Alone in Patients With Resectable Hepatocellular Carcinoma Beyond Milan Criteria
Brief Title: Neoadjuvant HAIC for Resectable Hepatocellular Carcinoma Beyond Milan Criteria
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Ming Shi, Proffessor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HCC-180302
Record Dates: First submitted 2018-03-11; First posted 2018-03-19 (Actual); Last update posted 2018-08-02 (Actual); Status verified 2018-07

CONDITIONS: Hepatocellular Carcinoma
Keywords: Neoadjuvant hepatic arterial infusion chemotherapy; BCLC A/B; FOLFOX; Resection
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Folfox protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Resection plus HAIC with FOLFOX (Experimental): Patients receive 4 times of neoadjuvant hepatic arterial infusion chemotherapy with FOLFOX and hepatic resection
  Interventions: Drug: FOLFOX; Procedure: Hepatic resection
- Resection (Active Comparator): Patients receive hepatic resection without neoadjuvant hepatic arterial infusion chemotherapy
  Interventions: Procedure: Hepatic resection

INTERVENTIONS:
Drug: FOLFOX — Hepatic intra-arterial infusion via the tumor feeding arteries of Oxaliplatin , fluorouracil, and leucovorin
  Other Names: Hepatic Arterial Infusion Chemotherapy of FOLFOX
  Arms: Resection plus HAIC with FOLFOX
Procedure: Hepatic resection — R0 resection

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of resection plus neoadjuvant hepatic arterial infusion chemotherapy (HAIC) compared with resection alone in patients with resectable hepatocellular carcinoma beyond Milan criteria.

DETAILED DESCRIPTION:
Resection is the long-term therapeutic option for resectable hepatocellular carcinoma (HCC) patients. While a number of studies demonstrate poor effect and high relapse rate of resection for patients with resectable hepatocellular carcinoma beyond Milan criteria. Our previous prospective study also revealed that neoadjuvant transarterial chemoembolization (TACE) seems to confer a survival benefit for resectable HCC. Recently, the results of our previous prospective study suggested that, compared with TACE, hepatic arterial infusion chemotherapy (HAIC) may improve the survivals for HCC with large HCC.Thus, the investigators carried out this prospective randomized control to demonstrate the superiority of resection plus neoadjuvant HAIC over resection alone.

ELIGIBILITY:
Inclusion Criteria:

* The diagnosis of HCC was based on the diagnostic criteria for HCC used by the European Association for the Study of the Liver (EASL;
* Tumor burden beyond Milan criteria
* Diagnosed as resectable with consensus by the panel of liver surgery experts;
* No past history of resection, radiofrequency ablation, TACE, TAI, chemotherapy or molecule-targeted treatment;
* No Cirrhosis or cirrhotic status of Child-Pugh class A only;
* Meet the following laboratory parameters:(a) Platelet count ≥ 75,000/μL; (b)Hemoglobin ≥ 8.5 g/dL;(c) Total bilirubin ≤ 30mmol/L;(d) Serum albumin

  ≥ 32 g/L;(e) ASL and AST ≤ 6 x upper limit of normal;(f) Serum creatinine

  ≤ 1.5 x upper limit of normal;(g) INR > 2.3 or PT/APTT within normal limits; (h) Absolute neutrophil count (ANC) >1,500/mm3;
* Ability to understand the protocol and to agree to and sign a written informed consent document. Exclusion Criteria;
* Patients with clinically significant gastrointestinal bleeding within 30 days prior to study entry.
* Known of serious heart disease which can nor endure the treatment such as cardiac ventricular arrhythmias requiring anti-arrhythmic therapy
* Evidence of hepatic decompensation including ascites, gastrointestinal bleeding or hepatic encephalopathy
* Known history of HIV
* History of organ allograft
* Known or suspected allergy to the investigational agents or any agent given in association with this trial.
* Evidence of bleeding diathesis.
* Any other hemorrhage/bleeding event > CTCAE Grade 3
* Serious non-healing wound, ulcer, or bone fracture
* Known central nervous system tumors including metastatic brain disease
* Poor compliance that can not comply with the course of treatment and follow up.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 252 (Estimated)
Dates: Start 2018-03-02 (Actual); Primary Completion 2023-03-02 (Estimated); Study Completion 2023-03-02 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 60 months
  Time to death

SECONDARY OUTCOMES:
Disease-free survival | 60 months
  Time to recurrence or death
Adverse Events | 30 days
  Number of adverse events. Postoperative adverse events were graded based on CTCAE v4.0

CONTACTS AND LOCATIONS:
Overall Officials: Ming Shi, MD, Principal Investigator — The Department of Hepatobiliary Oncology of Sun Yat-sen University Cancer
Locations (7):
- China (7):
  - Dongguan People's Hospital, Dongguan, Guangdong
  - Cancer Center Sun Yat-sen University, Guangzhou, Guangdong
  - The First Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong
  - Guangzhou Twelfth People's Hospital, Guangzhou, Guangdong
  - Kaiping Central Hospital, Kaiping, Guangdong
  - The First Affiliated Hospital of University Of South China, Hengyang, Hunan
  - First Affiliated Hospital Of Xi'an Jiaotong University, Xi’an, Shanxi

IPD SHARING:
Plan to Share IPD: Undecided